CLINICAL TRIAL: NCT02323698
Title: The Effects of Intermittent Hypoxia on Leg Function in Human Spinal Cord Injury (Caffeine Substudy)
Brief Title: Effects of Caffeine and Intermittent Hypoxia on Leg Function in Human Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Randy Trumbower, PT, PhD, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P001940b; 5R01HD081274 (NIH)
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries
Keywords: hypoxia; spinal cord injury; rehabilitation; strength; walk; function; low oxygen
MeSH Terms: conditions — Spinal Cord Injuries; Hypoxia | interventions — Caffeine; Insemination, Artificial, Homologous; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Balanced design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caffeine/AIH (Active Comparator): Subjects with chronic, motor-incomplete SCI receive Caffeine then AIH
  Interventions: Drug: Caffeine; Other: AIH
- Placebo/AIH (Active Comparator): Subjects with chronic, motor-incomplete SCI receive Placebo then AIH
  Interventions: Other: AIH; Other: Placebo
- Caffeine/SHAM (Active Comparator): Subjects with chronic, motor-incomplete SCI receive Caffeine then SHAM
  Interventions: Drug: Caffeine; Other: SHAM

INTERVENTIONS:
Drug: Caffeine — Subjects will ingest capsules containing caffeine (up to 6mg/kg). Experiments will begin 30min after consumption to approximately coincide with peak plasma concentrations.Throughout the 30min wait time and experimentation, blood pressure and heart rate will be monitored.
  Other Names: caffeine anhydrous
  Arms: Caffeine/AIH; Caffeine/SHAM
Other: AIH — Participants will breathe intermittent low oxygen via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.10±0.02 (hypoxia). Throughout experimentation, blood pressure and heart rate will be monitored.
  Other Names: Acute intermittent hypoxia
  Arms: Caffeine/AIH; Placebo/AIH
Other: Placebo — This is a placebo counterpart to the caffeine drug. Subjects will ingest capsules containing dextrose. Experiments will begin 30min after consumption to mimic the caffeine drug protocol. Throughout experimentation, blood oxygenation, blood pressure and heart rate will be monitored.
  Arms: Placebo/AIH
Other: SHAM — This is a placebo counterpart to breathing intermittent low oxygen. Participants will breathe intermittent room air via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.21±0.02 (normoxia). Throughout experimentation, blood pressure and heart rate will be monitored.
  Arms: Caffeine/SHAM

SUMMARY:
Accumulating evidence suggests that repeatedly breathing low oxygen levels for brief periods (termed intermittent hypoxia) is a safe and effective treatment strategy to promote meaningful functional recovery in persons with chronic spinal cord injury (SCI). The goal of the study is to understand how caffeine may augment the effects of intermittent hypoxia on motor function and spinal plasticity (ability of the nervous system to strengthen neural pathways based on new experiences) following SCI.

DETAILED DESCRIPTION:
The investigators will examine the effects of acute intermittent hypoxia (AIH) as a possible therapeutic intervention to promote functionally useful motor recovery. In this sub-study, the investigators will assess changes in leg motor function in response to repetitive AIH with and without caffeine.

Participants will receive caffeine+AIH, placebo+AIH, caffeine+SHAM in a randomized order. Before each intervention round, subjects will be asked to avoid caffeine-containing substances for 48 hrs (> 5* half-life of ~7 hrs) prior to arrival to control for baseline plasma levels of caffeine. Subjects will then ingest capsules containing either placebo (dextrose) or caffeine (up to 6mg/kg). Capsules will be prepared by Johnson Compounding & Wellness. Blood samples will be collected before and after the breathing intervention to assess caffeine concentrations within the body.

During and after each intervention, both the rate and extent of magnitude changes in voluntary and involuntary muscle response behaviors important for walking will be compared between interventions within participants. Repeated measurements will be collected on all subjects that participate in the multiple interventions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and 75 years (the latter to reduce likelihood of heart disease)
* medical clearance to participate
* lesion at or below C2 and above L5 with non-progressive etiology
* classified as motor-incomplete with visible volitional leg movement
* injury greater than 6 months
* ability to advance one step overground without human assistance

Exclusion Criteria:

* Concurrent severe medical illness (i.e., infection, cardiovascular disease, ossification, recurrent autonomic dysreflexia, unhealed decubiti, and history of pulmonary complications)
* Pregnant women because of the unknown affects of AIH on pregnant women and fetus
* History of seizures, brain injury, and/or epilepsy
* Undergoing concurrent physical therapy
* Diabetes
* Cirrhosis
* Caffeine and/or NSAID allergies or intolerances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Trumbower, PT, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trumbower RD. Stimulating the Injured Spinal Cord: Plenty to Grasp. J Neurotrauma. 2018 Sep 15;35(18):2143-2144. doi: 10.1089/neu.2018.5993. No abstract available. PMID 30009669
- [Background] Sohn WJ, Tan AQ, Hayes HB, Pochiraju S, Deffeyes J, Trumbower RD. Variability of Leg Kinematics during Overground Walking in Persons with Chronic Incomplete Spinal Cord Injury. J Neurotrauma. 2018 Nov 1;35(21):2519-2529. doi: 10.1089/neu.2017.5538. Epub 2018 Jun 5. PMID 29648987
- [Background] Trumbower RD, Hayes HB, Mitchell GS, Wolf SL, Stahl VA. Effects of acute intermittent hypoxia on hand use after spinal cord trauma: A preliminary study. Neurology. 2017 Oct 31;89(18):1904-1907. doi: 10.1212/WNL.0000000000004596. Epub 2017 Sep 29. PMID 28972191
- [Background] Peters DM, Thibaudier Y, Deffeyes JE, Baer GT, Hayes HB, Trumbower RD. Constraints on Stance-Phase Force Production during Overground Walking in Persons with Chronic Incomplete Spinal Cord Injury. J Neurotrauma. 2018 Feb 1;35(3):467-477. doi: 10.1089/neu.2017.5146. Epub 2017 Oct 27. PMID 28762876
- [Background] Hayes HB, Chvatal SA, French MA, Ting LH, Trumbower RD. Neuromuscular constraints on muscle coordination during overground walking in persons with chronic incomplete spinal cord injury. Clin Neurophysiol. 2014 Oct;125(10):2024-35. doi: 10.1016/j.clinph.2014.02.001. Epub 2014 Feb 14. PMID 24618214
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- See also: INSPIRE Lab Website — http://inspire-lab.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Caffeine/AIH First, Then Placebo/AIH, Then Caffeine/SHAM; Placebo/AIH First, Then Caffeine/AIH, Then Caffeine/SHAM; Caffeine/SHAM First, Then Caffeine/AIH, Then Placebo/AIH; Caffeine/AIH First, Then Caffeine/SHAM, Then Placebo/AIH; Placebo/AIH First, Then Caffeine/SHAM, Then Caffeine/AIH; Caffeine/SHAM First, Then Placebo/AIH, Then Caffeine/AIH: Subjects ingest Caffeine/Placebo 30 minutes prior to AIH/SHAM breathing intervention in this cross-over study. All participants are assigned to receive all three intervention combinations of Caffeine/AIH, Placebo/AIH, and Caffeine/SHAM in a randomized order with each intervention lasting 5 days followed by 14 days of washout prior to starting the next intervention. Throughout experimentation, blood oxygenation, blood pressure and heart rate are monitored.
  Caffeine: Subjects ingest capsules containing caffeine (up to 6mg/kg). Breathing intervention begins 30min after consumption to approximately coincide with peak plasma concentrations.
  Placebo: This is a placebo counterpart to the caffeine drug. Subjects ingest capsules containing dextrose. Breathing intervention begins 30min after consumption to mimic the caffeine drug protocol.
  AIH: Participants breathe intermittent low oxygen via air generators. The generators fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration is continuously monitored to ensure intermittent delivery of FIO2 (fraction of inspired oxygen) = 0.10±0.02 (hypoxia) at 1-minute intervals.
  SHAM: This is a placebo counterpart to breathing intermittent low oxygen. Participants breathe intermittent room air via air generators. The generators fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration is continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.21±0.02 (normoxia).
Period: Overall Study
Arm/Group | Caffeine/AIH First, Then Placebo/AIH, Then Caffeine/SHAM | Placebo/AIH First, Then Caffeine/AIH, Then Caffeine/SHAM | Caffeine/SHAM First, Then Caffeine/AIH, Then Placebo/AIH | Caffeine/AIH First, Then Caffeine/SHAM, Then Placebo/AIH | Placebo/AIH First, Then Caffeine/SHAM, Then Caffeine/AIH | Caffeine/SHAM First, Then Placebo/AIH, Then Caffeine/AIH
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed First Intervention (5 Days) | 2 | 2 | 2 | 2 | 2 | 2
Completed Second Intervention (5 Days) | 2 | 2 | 1 | 2 | 2 | 2
Completed Third Intervention (5 Days) | 2 | 2 | 0 | 2 | 1 | 2
Completed | 2 | 2 | 0 | 2 | 1 | 2
Not Completed | 0 | 0 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects ingest Caffeine/Placebo 30 minutes prior to AIH/SHAM breathing intervention in this cross-over study. All participants are assigned to receive all three intervention combinations of Caffeine/AIH, Placebo/AIH, and Caffeine/SHAM in a randomized order with each intervention lasting 5 days followed by 14 days of washout prior to starting the next intervention. Throughout experimentation, blood oxygenation, blood pressure and heart rate are monitored.
  Caffeine: Subjects ingest capsules containing caffeine (up to 6mg/kg). Breathing intervention begins 30min after consumption to approximately coincide with peak plasma concentrations.
  Placebo: This is a placebo counterpart to the caffeine drug. Subjects ingest capsules containing dextrose. Breathing intervention begins 30min after consumption to mimic the caffeine drug protocol.
  AIH: Participants breathe intermittent low oxygen via air generators. The generators fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration is continuously monitored to ensure intermittent delivery of FIO2 (fraction of inspired oxygen) = 0.10±0.02 (hypoxia) at 1-minute intervals.
  SHAM: This is a placebo counterpart to breathing intermittent low oxygen. Participants breathe intermittent room air via air generators. The generators fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration is continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.21±0.02 (normoxia).
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants with Level of Spinal Cord Injury (C2-L5) [Number; unit: Participants] | 10
Time Since Injury [Mean (Standard Deviation); unit: years] | 8 (12)
CYP1A2*1F SNP [Number; unit: participants] — Participant genotype for CYP1A2 polymorphism was assessed. Homozygosity for A/A is considered a fast metabolizer of caffeine and C/A heterozygosity is considered a slow metabolizer of caffeine.
  participants
    A/A | 3
    C/A | 8
10 Meter Walk Test [Mean (Standard Deviation); unit: Seconds] — Speed will be assessed using the time required to walk 10 meters (10MWT).
  Seconds | 32.8 (31.0)

OUTCOME MEASURES:

1. Primary Outcome: 10 Meter Walk Time
Description: Speed will be assessed using the time required to walk 10 meters (10MWT) relative to baseline.
Time Frame: Baseline, after intervention (day 5), and at follow-ups (one week and two weeks)
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Caffeine/AIH | Placebo/AIH | Caffeine/SHAM
Number analyzed (Participants) | 10 | 7 | 10
Seconds
  Day 5 (Relative to Baseline) | -5.0 (2.2) | -4.9 (2.2) | -4.6 (2.1)
  Day 12 (Relative to Baseline) | -5.5 (2.7) | -1.7 (1.3) | 0.9 (1.5)
  Day 19 (Relative to Baseline) | -6.5 (3.3) | 0.4 (2.6) | -0.1 (0.6)

2. Secondary Outcome: 6 Minute Walk Test
Description: Measure participant's distance walked in 6 minutes (meters).
Time Frame: Baseline, after intervention (day 5), and at follow-ups (one week and two weeks)
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Caffeine/AIH | Placebo/AIH | Caffeine/SHAM
Number analyzed (Participants) | 11 | 12 | 8
Meters
  Day 5 (Relative to Baseline) | 24.1 (8.3) | 17.1 (7.3) | 6.2 (8.7)
  Day 12 (Relative to Baseline) | 23.7 (7.7) | 15.7 (7.3) | 9.2 (9.3)
  Day 19 (Relative to Baseline) | 22.4 (8.0) | 24.2 (7.6) | -2.7 (8.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Caffeine/AIH | Placebo/AIH | Caffeine/SHAM
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT02323698/Prot_SAP_000.pdf